CLINICAL TRIAL: NCT02072954
Title: A Multicentric, Open Label, Randomized, Balanced, Two Treatment, Three Period, Three Sequence, Crossover, Multiple Dose, Steady State Bioequivalence Study of Asenapine Sublingual Tablets, 10 mg Manufactured by AMNEAL PHARMACEUTICALS, USA With Reference Product SAPHRIS® (Asenapine) Sublingual Tablets, 10 mg Manufactured by Catalent UK Swindon Zydis Ltd., Blagrove, Swindon, Wiltshire, SN5 8RU, UK; Distributed by Merck Sharp & Dohme Corp., a Subsidiary of Merck & Co., Inc., Whitehouse Station, NJ, 08889, USA in Adult Human Male & Female Patients Under Fasting Condition.
Brief Title: Bioequivalence Fasting Study in Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amneal Pharmaceuticals, LLC (Industry)
Collaborators: Accutest Research Laboratories (I) Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARL/CT/13/003; CTRI No. CTRI/2013/11/004152 (Other: Clinical Trials Registration India)
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asenapine Sublingual Tablets (Experimental): Asenapine Sublingual Tablets, 10 mg. Twice daily for a period of 7 days
  Interventions: Drug: Asenapine Sublingual Tablets 10 mg
- Saphris Subligual Tablets (Active Comparator): Asenapine Sublingual Tablets, 10 mg. Twice daily for 2 periods of 7 days each.
  Interventions: Drug: Asenapine Sublingual Tablets 10 mg

INTERVENTIONS:
Drug: Asenapine Sublingual Tablets 10 mg — White to off-white, round, uncoated,unscored, flat-faced radius edge tablet. Debossed with A on one side and 17 on the other side
  Arms: Asenapine Sublingual Tablets
Drug: Asenapine Sublingual Tablets 10 mg — Round, white to off-white sublingual tablets, with "10" on one side within a circle
  Arms: Saphris Subligual Tablets

SUMMARY:
To compare and evaluate the oral bioavailability of Asenapine Sublingual Tablets, 10 mg manufactured by AMNEAL PHARMACEUTICALS, USA with SAPHRIS® (asenapine) sublingual tablets, 10 mg.

DETAILED DESCRIPTION:
To compare and evaluate the oral bioavailability of Asenapine Sublingual Tablets, 10 mg manufactured by AMNEAL PHARMACEUTICALS, USA with SAPHRIS® (asenapine) sublingual tablets, 10 mg following a multiple-dose administration in adult human patients who are receiving a stable twice daily dose of asenapine maleate EQ 10 mg base.

To monitor the safety and tolerability of a multiple doses of asenapine sublingual tablets 10 mg in adult human patients who are receiving a stable twice daily dose of asenapine maleate EQ 10 mg base.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex with age between 18 to 65 years (both inclusive) and have been taking a stable dose of asenapine maleate sublingual tablet, EQ 10 mg base twice daily therapy for at least three months.
* Willing and able to comply with study visit schedule and other protocol requirements as indicated by signed written informed consent witnessed by a legally acceptable representative.
* Females of childbearing (who has not completed 01 year after menopause & have not gone through hysterectomy or bilateral tubal ligation) potential must have a negative pregnancy test (at screening, before randomization and before check-in to housing) as well as must be non-lactating at screening and must agree to use an effective contraceptive method during study.

Exclusion Criteria:

* History of allergic or adverse reactions to asenapine maleate or olanzapine as judged by investigator
* If consuming tobacco orally (spit tobacco, gutka, pan masala, pan, etc.)
* A history of severe hepatic impairment, drug induced leukopenia/ neutropenia, congenital prolongation of the QT interval, cardiac arrhythmias, myocardial infarction or unstable heart disease
* Concurrent primary psychiatric or neurological diagnosis, including organic mental disorder, severe tardive dyskinesia, or idiopathic Parkinson's disease
* Abnormal laboratory results
* A history of granulocytopenia or myeloproliferative disorders (drug-induced or idiopathic)
* A medical or surgical condition that might interfere with the absorption, metabolism, or excretion of asenapine maleate
* History of multiple syncopal episodes
* History of epilepsy or risk for seizures
* Any condition/ Abnormal baseline findings that in the investigators' judgment might increase the risk to the patient (e.g. Significant orthostatic hypotension defined as a drop in systolic blood pressure of 30 mm Hg or more and/or a drop in diastolic blood pressure of 20 mm Hg or more on standing) or decrease the chance of obtaining satisfactory data needed to obtain the objective of the study.
* A history of alcohol or drug dependence by DSM-IV criteria during the 6-month period immediately prior to study entry
* Positive tests for drug or alcohol abuse at screening or baseline
* Use of any of the following medication in the 14 days preceding enrollment: Strong CYP3A4 inhibitors, Strong CYP3A4 inducers, CYP1A2 inhibitors, Antihypertensive medication or any medication that might predispose to orthostatic hypotension, Drugs known to suppress bone marrow function, medications known to prolong the QTc interval.
* Participation in any other clinical study or receipt of treatment with any investigational drug or device within 1 month prior Screening.
* Blood donation/ loss exceeding 550 mL within last 90 days.
* Any expected changes in concomitant medications during the period of study
* Compliance with outpatient medication schedule not expected

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
AUC 0-tau | Dosing interval on day 7
  The area under plasma concentration versus time curve, over the steady state dosing interval, calculated using linear trapezoidal method.
Cmax | Dosing interval on day 7
  Maximum measured plasma concentration over the steady state doing interval

SECONDARY OUTCOMES:
Cmin | Dosing interval on day 7
  Minimum measured plasma concentration over the steady state dosing interval
Tmax | Dosing interval on day 7
  Time the maximum measured plasma concentration over the steady state dosing interval
Cavg | Dosing interval on day 7
  Average calculated plasma concentration over the steady state dosing interval
Percentage Fluctuation | Dosing interval on day 7
  [Cmax - Cmin/ Cavg] x 100

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh Jani, MD, Principal Investigator — Accutest Reserach laboratories (i) Pvt. Ltd.
Locations (2):
- India (2):
  - Shri Hatkesh Healthcare Foundation, Jūnāgadh, Gujurat
  - Divyam Hospital, Surat, Gujurat